CLINICAL TRIAL: NCT05803096
Title: Self-Administered Nitrous Oxide (SANO) During Transrectal Prostate Biopsy to Reduce Patient Anxiety and Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Heidi Rayala, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021P-000715
Record Dates: First submitted 2023-02-28; First posted 2023-04-07 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Prostate Disease; Malignancy; Benign Prostatic Hyperplasia; Prostate Cancer; Prostate Adenocarcinoma; Anxiety and Fear; Pain
Keywords: prostate biopsy; nitrous oxide; prostate cancer; ambulatory; patient experience of care
MeSH Terms: conditions — Prostatic Diseases; Neoplasms; Prostatic Hyperplasia; Prostatic Neoplasms; Anxiety Disorders; Pain | interventions — Nitrous Oxide; Oxygen

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to either SANO (treatment) or oxygen (placebo control) after completion of baseline assessment. The results of the randomization will not be disclosed to patients as part of the study (patient-blinded).
Who Masked: Participant, Care Provider
Masking Description: The operating urologist and study participant will be blinded to group assignment for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-Administered Nitrous Oxide (Active Comparator): Patients will receive SANO in addition to periprostatic bupivacaine nerve block for the duration of prostate biopsy.
  After the Urologist describes the procedure, the SANO group will have nitrous oxide turned on to 30%, ensuring that the patient is relaxed but still conversant through the procedure. The nitrous will be adjust up or down based on the patient's response to the question "are you feeling the nitrous" and "are you happy at this level". The range will be between 25 - 45%. At the end of the procedure, the SANO group will be turned down to 0% nitrous oxide, and 100% oxygen will be administered through the mask for an additional 2-3 minutes as the patient is cleaned up and repositioned to the supine position.
  Interventions: Drug: Self-Administered Nitrous Oxide
- Oxygen (Placebo Comparator): Patients will receive 100% oxygen at 10 Liters/minute for the duration of prostate biopsy.
  Interventions: Other: Oxygen

INTERVENTIONS:
Drug: Self-Administered Nitrous Oxide — Nitrous oxide administered at concentrations of mild sedation (20-45%) for the duration of prostate biopsy.
  Other Names: nitrous oxide
  Arms: Self-Administered Nitrous Oxide
Other: Oxygen — Oxygen will be administered at 10 Liters/min for the duration of prostate biopsy.
  Arms: Oxygen

SUMMARY:
Transrectal prostate biopsy is a commonly performed ambulatory procedure for diagnosing prostate cancer. Prostate biopsy are associated with pain or anxiety. Nitrous oxide (or laughing gas) is a well-known inhaled anesthetic which is frequently used in dental offices and for pediatric procedures to alleviate a patient's anxiety and pain. This study seeks to determine whether administration of nitrous oxide at the time of prostate biopsy will improve a patient's experience of care.

DETAILED DESCRIPTION:
Nitrous oxide is a well-tolerated inhaled anesthetic that has been used for decades in pediatric and adult populations and is largely viewed as effective and safe. In addition to analgesic effect, nitrous oxide also produces a dissociative euphoria and amnesia that could potentially improve patients' anxiety and experience of cancer care. When used as a single agent at concentrations ≤50%, the American Society of Anesthesiologists (ASA) classifies nitrous oxide as Minimal Sedation, producing a state in which a patient responds normally to verbal commands, maintains airway reflexes, and spontaneous ventilation. Over the past several decades nitrous oxide has become less common due to concerns of nitrous oxide environmental exposure to the care team. There are now Federal Drug Administration (FDA)-approved systems that allow patient self-administered nitrous oxide (SANO), and importantly, include a scavenger system to eliminate exhaled environmental nitrous oxide. These systems are rapidly being adopted throughout the United States in Urology practices, but to date, there have been no studies evaluating patient outcomes and possible risks with the adjunct use of SANO. This study is a prospective, randomized, controlled trial to assess patient perceived pain and anxiety related to prostate needle biopsy with or without SANO, and the frequency of complications associated with SANO. A secondary aim will be to demonstrate that the SANO at the time of prostate biopsy does not significantly increase burden on Urologist productivity, nor increase the difficulty of operator ease in performing the prostate needle biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Biological male
* Aged 18 to 85 years
* Scheduled for clinically-indicated prostate needle biopsy
* Suitable for nitrous oxide/oxygen with willingness to be randomized to inhaled SANO or inhaled oxygen during the procedure
* Access to an email and computer

Exclusion Criteria:

* Perioral facial hair impeding good mask seal
* Learning disabilities and/or inability to cognitively complete survey questions
* Taken a pre-procedure benzodiazepine or narcotic.
* Has any of the following medical conditions:

  1. Inner ear, bariatric or eye surgery within the last 2 weeks,
  2. Current emphysematous blebs,
  3. Severe B-12 deficiency.
  4. Bleomycin chemotherapy within the past year.
  5. Class III or higher heart failure.
  6. Undergoing novel therapy for prostate cancer

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants with a prostate may be eligible for the study.
Enrollment: 143 (Actual)
Dates: Start 2021-12-12 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Rayala, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
IPD is not intended to be shared to personnel outside of pre-defined research staff.

REFERENCES:
- [Background] Loeb S, Carter HB, Berndt SI, Ricker W, Schaeffer EM. Complications after prostate biopsy: data from SEER-Medicare. J Urol. 2011 Nov;186(5):1830-4. doi: 10.1016/j.juro.2011.06.057. Epub 2011 Sep 23. PMID 21944136
- [Background] Rosario DJ, Lane JA, Metcalfe C, Donovan JL, Doble A, Goodwin L, Davis M, Catto JW, Avery K, Neal DE, Hamdy FC. Short term outcomes of prostate biopsy in men tested for cancer by prostate specific antigen: prospective evaluation within ProtecT study. BMJ. 2012 Jan 9;344:d7894. doi: 10.1136/bmj.d7894. PMID 22232535
- [Background] Jastak JT, Donaldson D. Nitrous oxide. Anesth Prog. 1991 Jul-Oct;38(4-5):142-53. No abstract available. PMID 1819967
- [Background] Practice Guidelines for Moderate Procedural Sedation and Analgesia 2018: A Report by the American Society of Anesthesiologists Task Force on Moderate Procedural Sedation and Analgesia, the American Association of Oral and Maxillofacial Surgeons, American College of Radiology, American Dental Association, American Society of Dentist Anesthesiologists, and Society of Interventional Radiology. Anesthesiology. 2018 Mar;128(3):437-479. doi: 10.1097/ALN.0000000000002043. No abstract available. PMID 29334501

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of note, 143 patients were consented for procedure, but only 133 were randomized. This discrepancy was due to study staff availability or patient cancellation of procedure.
Groups:
- Self-Administered Nitrous Oxide: Patients will receive SANO in addition to periprostatic bupivacaine nerve block for the duration of prostate biopsy.
  After the Urologist describes the procedure, the SANO group will have nitrous oxide turned on to 30%, ensuring that the patient is relaxed but still conversant through the procedure. The nitrous will be adjust up or down based on the patient's response to the question "are you feeling the nitrous" and "are you happy at this level". The range will be between 25 - 45%. At the end of the procedure, the SANO group will be turned down to 0% nitrous oxide, and 100% oxygen will be administered through the mask for an additional 2-3 minutes as the patient is cleaned up and repositioned to the supine position.
  Self-Administered Nitrous Oxide: Nitrous oxide administered at concentrations of mild sedation (20-45%) for the duration of prostate biopsy.
Period: Overall Study
Arm/Group | Self-Administered Nitrous Oxide | Oxygen
Started | 66 | 67
Completed | 61 | 67
Not Completed | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-Administered Nitrous Oxide | Oxygen | Total
Number analyzed (Participants) | 61 | 67 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (11.5) | 65.8 (7.8) | 65.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 61 | 67 | 128
Race/Ethnicity, Customized [Number; unit: participants]
  White | 50 | 56 | 106
  Black/African American | 8 | 9 | 17
  Other | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61 | 67 | 128
History of Prostate Cancer Prior to Enrollment [Count of Participants; unit: Participants] | 26 | 17 | 43
Past Medical History of Depression [Count of Participants; unit: Participants] | 7 | 10 | 17
Past Medical History of Anxiety [Count of Participants; unit: Participants] | 10 | 10 | 20
Pre-Biopsy VAS-Anxiety [Median (Inter-Quartile Range); unit: units on a scale] — Pre-procedural anxiety was assessed using the Visual Analog Scale for Anxiety (VAS-A, range:0-10, higher scores indicating worse anxiety).
  units on a scale | 3 [0 to 5] | 2 [0 to 5] | 2 [0 to 5]
Pre-Biopsy VAS-Pain [Median (Inter-Quartile Range); unit: units on a scale] — Pre-procedural pain was measured by the Visual Analog Scale for Pain (VAS-P, range:0-10, with greater scores indicating worse pain).
  units on a scale | 0 [0 to 1] | 0 [0 to 0] | 0 [0 to 0]
Pre-Biopsy STAI [Median (Inter-Quartile Range); unit: units on a scale] — Pre-procedural anxiety was assessed using the State Trait Anxiety Inventory (STAI, range:6-24, higher scores indicate worse anxiety)
  units on a scale | 12 [9 to 15] | 12 [8 to 14] | 12 [8 to 14]

OUTCOME MEASURES:

1. Primary Outcome: Post-biopsy Pain (VAS-P)
Description: Pain experienced immediately following prostate biopsy as measured by a Visual Analog Scale for Pain (VAS-P) (range: 0 [no pain] - 10 [worst pain])
Time Frame: 5-minutes after prostate biopsy
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Self-Administered Nitrous Oxide | Oxygen
Number analyzed (Participants) | 61 | 67
score on a scale | 1 [0 to 2] | 1 [0 to 2]

2. Primary Outcome: Post-biopsy Anxiety (VAS-A)
Description: Anxiety experienced immediately following prostate biopsy as measured by a Visual Analog Scale for Anxiety (VAS-A) (range: 0 [no anxiety] - 10 [worst anxiety])
Time Frame: 5-minutes after prostate biopsy
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Self-Administered Nitrous Oxide | Oxygen
Number analyzed (Participants) | 61 | 67
score on a scale | 0 [0 to 3] | 1 [0 to 3]

3. Primary Outcome: Post-biopsy Anxiety Traits (STAI)
Description: Anxious traits exhibited after prostate biopsy as measured by the State Trait Anxiety Inventory (STAI) (range: 6-36; 36 being 'worst' anxiety).
Time Frame: 5-minutes after prostate biopsy
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Self-Administered Nitrous Oxide | Oxygen
Number analyzed (Participants) | 61 | 67
score on a scale | 11 [7 to 14] | 12 [9 to 14]

4. Secondary Outcome: Time of Prostate Biopsy
Description: Length of procedure will be compared between arms to assess whether SANO significantly lengthens prostate biopsy
Time Frame: Length of prostate biopsy; up to 30 minutes
Measure: Mean (Inter-Quartile Range); unit: minutes
Arm/Group | Self-Administered Nitrous Oxide | Oxygen
Number analyzed (Participants) | 61 | 67
minutes | 10.6 [9 to 12.6] | 10.3 [8.5 to 11.9]

5. Secondary Outcome: Operator Assessment of "Tolerating Insertion of Rectal Probe"
Description: Operating urologist filled out a survey to assess their perception of patient: Tolerating Insertion of rectal probe. Responses were scored on a 3-point Likert scale as 1 (worse than expected), 2 (as expected), or 3 (better than expected).
Time Frame: Immediately after prostate biopsy; within 5 minutes after completion of biopsy.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Self-Administered Nitrous Oxide | Oxygen
Number analyzed (Participants) | 61 | 67
score on a scale | 2 [2 to 3] | 2 [2 to 3]

6. Secondary Outcome: Operator Assessment of "Patient Maintenance of Positioning"
Description: Operating urologist filled out a survey to assess their perception of patient: Patient maintenance of positioning. Responses were scored on a 3-point Likert scale as 1 (worse than expected), 2 (as expected), or 3 (better than expected).
Time Frame: Immediately after prostate biopsy; within 5 minutes after completion of biopsy.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Self-Administered Nitrous Oxide | Oxygen
Number analyzed (Participants) | 61 | 67
score on a scale | 2 [2 to 3] | 2 [2 to 3]

7. Secondary Outcome: Operator Assessment of "Patient Tolerance of Procedure"
Description: Operating urologist filled out a survey to assess their perception of patient: Patient Tolerance of Procedure. Responses were scored on a 3-point Likert scale as 1 (worse than expected), 2 (as expected), or 3 (better than expected).
Time Frame: Immediately after prostate biopsy; within 5 minutes after completion of biopsy.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Self-Administered Nitrous Oxide | Oxygen
Number analyzed (Participants) | 61 | 67
score on a scale | 2 [2 to 3] | 2 [2 to 3]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Self-Administered Nitrous Oxide | Oxygen
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/67
Other Adverse Events (participants affected / at risk) | 1/61 | 2/67
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self-Administered Nitrous Oxide (N=61) | Oxygen (N=67)
Facial Flushing (General disorders) | 1 (1) | 0 (0) — Facial Flushing during procedure
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1) — Urinary Retention with need for catheter
Acute Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) — Acute Cholangitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT05803096/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT05803096/ICF_000.pdf